CLINICAL TRIAL: NCT05644938
Title: Optimizing Door-to-reperfusion Times of One-stop Management in Acute Ischemic Stroke Trial
Brief Title: Optimizing Door-to-reperfusion Times of One-stop Management in Acute Ischemic Stroke
Acronym: ORETOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Can Tho Stroke International Services Hospital (Other)
Collaborators: Siemens Healthineers AG (Unknown)
Responsible Party: Principal Investigator, Dr. Cuong Tran Chi, Principal Investigator, Can Tho Stroke International Services Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CanTho SIS Hospital
Record Dates: First submitted 2022-11-26; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; angiosuite; reperfusion times; One-stop
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, single blind when patients are only blinded to the allocation, our clinical trial was conducted comparing One-stop (OS) management with our standard workflow (SW) in treatment of acute ischemic stroke from 12/2022 - 11/2023 at Can Tho SIS General Hospital. Patients were enrolled according to 1:1 enroll ratio (OS: SW). The OS group transferred directly to biplane flat panel detector computed tomography perfusion (FD-CTP) to consider recanalization by either intervention or recombinant Tissue Plasminogen Activator (rTPA) in the angiosuite, whereas the SW group was either transferred to angiosuite or received rTPA, if indicated, after the results of Magnetic resonance imaging (MRI) and Magnetic resonance angiography (MRA) at admission
Who Masked: Participant
Masking Description: Patients are only blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard workflow (SW) (Active Comparator): Acute ischemic stroke caused by large vessel occlusion was diagnosed by Magnetic resonance imaging (MRI) and Magnetic resonance angiography (MRA) at admission in MRI room + Recanalization therapy in angiosuite
  Interventions: Procedure: Standard workflow
- One-stop (OS) (Experimental): Acute ischemic stroke caused by large vessel occlusion was diagnosed + Recanalization therapy by the ﬂat-detector computed tomography in angiosuite at the same time.
  Interventions: Procedure: One-stop

INTERVENTIONS:
Procedure: Standard workflow — The SW group was either transferred to angiosuite or received rTPA, if indicated, after the results of Magnetic resonance imaging (MRI) and Magnetic resonance angiography (MRA) at admission.
  Other Names: SW
  Arms: Standard workflow (SW)
Procedure: One-stop — The OS group transferred directly to ﬂat-detector computed tomography to consider recanalization by either intervention or recombinant Tissue Plasminogen Activator (rTPA) in the angiosuite.
  Other Names: OS
  Arms: One-stop (OS)

SUMMARY:
Time is one of the most important in the decision of treatment of acute ischemic stroke. The optimal One-stop management from admission to recanalization associated with reduction of in-hospital times. The development of ﬂat-detector computed tomography perfusion capable angio-suite allowed One-stop management to be improved treatment time better and better. To compare One-stop management versus our standard workflow in shortening door-to-recanalization time.

DETAILED DESCRIPTION:
Acute ischemic stroke is one of the diseases associated with stroke onset time, especially in the case of large vessel occlusion within 6 hours. This is the reason why endovascular reperfusion therapy (mechanical thrombectomy, angioplasty, stent,…) is recommended to be performed as soon as possible in the comprehensive stroke centers. The successful recanalization within 6 hours demonstrated the efficacy that helps to improve the functional outcome by trials. Besides, the strategies shortening time from admission to successful recanalization are essential for the treatment of acute ischemic stroke due to large vessel occlusion. Nevertheless, the optimizing door-to-groin puncture and door to recanalization Time are the great challenge to benefit most patients with the endovascular therapy. In recent years, the One - stop management (direct transport to the angiosuite workflow) which means that the recanalization therapy is considered to perform immediately based on the diagnostic angiograms and perfusion maps relating to acute ischemic stroke caused by large vessel occlusion by the ﬂat-detector computed tomography at the angiosuite at the same time. We hypothesized that one-stop management is feasible and reduces more intrahospital time delays than our standard workflow previously published.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke in the anterior circulation caused by large vessel occlusion.
* National Institute of Health Stroke Scale (NIHSS) ≥10.
* Premorbid modified Rankin Scale (mRS) ≤ 2
* Target Mismatch profile: CBF < 30% volume < 100ml, Mismatch volume ≥ 15 ml and Mismatch Ratio >1.8.
* Available angiosuite.
* CBF < 30% volume: 70 - 100 ml when non-contrast computed tomography (NCCT) Alberta Stroke Program Early Computed Tomography Scores (ASPECTS) was 3 - 5 and/or beyond 6 hours after symptom onset

Exclusion Criteria:

* Evidence of intracranial tumors, the encephalitis, the hemorrhage: either an intracranial hemorrhage (ICH) or subarachnoid hemorrhage (SAH) by the biplane flat panel detector computed tomography.
* Participated in another studies.
* Loss to follow-up after discharge.
* A severe or fatal combined illness before acute stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Door-to-reperfusion times | 1 day (During intrahospital)
  Door-to-reperfusion times was defined as the time from admission in emergency department to recanalization in case of large vessel occlusion at the angiosuite..
Functional 3 - month outcome rate | 3 months after procedure
  Functional 3 - month outcome rate was accessed by modified Rankin Score (mRS), which comprised of included good (mRS 0 - ≤ 2) and fair (mRS 3).

CONTACTS AND LOCATIONS:
Overall Officials: Cuong C Tran, PhD, Study Director — Can Tho Stroke International Services General Hospital
Locations (1):
- Can Tho SIS Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Requena M, Olive-Gadea M, Muchada M, Hernandez D, Rubiera M, Boned S, Pinana C, Deck M, Garcia-Tornel A, Diaz-Silva H, Rodriguez-Villatoro N, Juega J, Rodriguez-Luna D, Pagola J, Molina C, Tomasello A, Ribo M. Direct to Angiography Suite Without Stopping for Computed Tomography Imaging for Patients With Acute Stroke: A Randomized Clinical Trial. JAMA Neurol. 2021 Sep 1;78(9):1099-1107. doi: 10.1001/jamaneurol.2021.2385. PMID 34338742
- [Result] Kurmann CC, Kaesmacher J, Cooke DL, Psychogios M, Weber J, Lopes DK, Albers GW, Mordasini P. Evaluation of time-resolved whole brain flat panel detector perfusion imaging using RAPID ANGIO in patients with acute stroke: comparison with CT perfusion imaging. J Neurointerv Surg. 2023 Apr;15(4):387-392. doi: 10.1136/neurintsurg-2021-018464. Epub 2022 Apr 8. PMID 35396333
- [Result] Brehm A, Tsogkas I, Maier IL, Eisenberg HJ, Yang P, Liu JM, Liman J, Psychogios MN. One-Stop Management with Perfusion for Transfer Patients with Stroke due to a Large-Vessel Occlusion: Feasibility and Effects on In-Hospital Times. AJNR Am J Neuroradiol. 2019 Aug;40(8):1330-1334. doi: 10.3174/ajnr.A6129. Epub 2019 Jul 11. PMID 31296523